CLINICAL TRIAL: NCT06880575
Title: Seniors Integrated Longitudinal cardioVascular Evaluation of Coronary Heart Disease: a Multicenter, Prospective Registry in China (SILVER-China)
Acronym: SILVER-China
Status: Recruiting | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Fusui Ji, MD, Chief physician and dean of Beijing Hospital, Beijing Hospital
Other Study IDs: BJ-2024-140; BJ-2024-140 (Other Grant/Funding Number: Central high-level hospital clinical scientific research business expenses special cohort special project)
Record Dates: First submitted 2025-03-14; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: Coronary Arterial Disease (CAD); ELDERLY PEOPLE
Keywords: Coronary Heart Disease; Chinese Elderly; Cohort Study
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elderly patients with coronary heart disease: 1. Establish a cohort and biological sample bank of elderly patients with coronary heart disease
  2. Establish a risk prediction model and clinical diagnosis and treatment optimization plan for elderly patients with coronary heart disease
  3. Systematically study the multi-dimensional feature spectrum of elderly patients with coronary heart disease

SUMMARY:
This study aims to establish a nationwide cohort and biobank of elderly patients with coronary heart disease (CHD) and to develop risk prediction models and clinical treatment optimization plans based on this data. The specific research content is as follows:

The Study plan to continuously enroll hospitalized elderly CHD patients across 50 centers nationwide. Using networked electronic data collection technology, standardized methods and protocols will be used to gather demographic information (such as age, gender, education level, income, etc.), clinical information (medical history, past treatment records, current treatment plans, surgical records, medication use, etc.), lifestyle information (dietary habits, exercise frequency, smoking, drinking, etc.), biological information (such as inflammatory markers, etc.), and physical examination data (such as blood pressure, ECG, sleep monitoring, imaging examinations, etc.). These patients will be followed up long-term (1 month, 6 months, 1 year, and annually thereafter for up to 5 years) to establish a database that meets international standards. Centers meeting the criteria will also retain biological samples, creating a multicenter biobank for elderly CHD patients.

Second, based on the established clinical cohort, a risk prediction model for elderly CHD patients will be developed, including mortality risk, ischemic risk, bleeding risk, etc. Additionally, optimized clinical diagnostic and treatment plans will be formulated to improve the treatment outcomes and quality of life for elderly CHD patients. This research is expected to provide scientific evidence and technical support for the prevention, diagnosis, and treatment of CHD in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

① Age requirements: Participants are ≥ 75 years old;

* This time he was admitted to the hospital due to angina pectoris and other coronary heart disease-related symptoms

  ③ Conform to the diagnosis of coronary heart disease: meet any one of the following conditions:
  1. This admission was performed for coronary angiography, coronary artery CTA confirmed coronary heart disease;
  2. Previous clear coronary angiography, coronary artery Coronary heart disease diagnosed by imaging evidence such as CTA evidence;
  3. The attending physician according to the patient's symptoms, medical history, myocardial injury markers, electrocardiogram, echo cardiography, myocardial radionuclide imaging, etc. diagnosed coronary heart disease.

     ④ Informed consent: Participants must be able to understand the content of the study, voluntarily participate in the study, and sign the informed consent form.

     Exclusion Criteria:
     * Combined with severe non-cardiovascular disease: life expectancy does not exceed 6 months, such as advanced cancer or other end-stage disease;
* Unable to cooperate with long-term follow-up: such as patients with severe cognitive impairment or severe mental illness; ③ Non-cardiogenic death within 24 hours after admission.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This project aims to establish a nationwide cohort of elderly patients with coronary heart disease. Elderly inpatients with coronary heart disease who met the admission criteria were selected into 50 centers across the country. To ensure the representativeness of the sample, the study will adopt the following strategies: extensive coverage of different regions: select medical institutions in major geographical regions of the country to ensure geographical diversity and regional representativeness of the data; Covering different types of medical institutions ensures that patients at different levels of medical services can be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10139 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | From enrollment to the end of follow up at 5 years
  MACCE, refers to the composite endpoint including all-cause mortality, non-fatal myocardial infarction, non-fatal stroke, and ischemia-driven revascularization

SECONDARY OUTCOMES:
all-cause mortality | From enrollment to the end of follow up at 5 years
cardiogenic death | From enrollment to the end of follow up at 5 years
non-fatal myocardial infarction | From enrollment to the end of follow up at 5 years
non-fatal stroke and ischemia-driven revascularization | From enrollment to the end of follow up at 5 years
stent thrombosis | From enrollment to the end of follow up at 5 years
major bleeding | From enrollment to the end of follow up at 5 years
  BARC type 3 and 5 bleeding
all BARC bleeding | From enrollment to the end of follow up at 5 years
NACE | From enrollment to the end of follow up at 5 years
  MACCE and major bleeding
Quality of life | From enrollment to the end of follow up at 5 years
  Smoking, alcohol consumption and nutrition were collected through questionnaires; Physical activity, sleep, and weakness were assessed by recognized scales such as the Physical Activity Scale for the Elderly (PASE), Epworth Lethargy Questionnaire, and FRAIL Weakness Scale; New York Heart Association (NYHA) cardiac function classification and Killip classification of acute myocardial infarction were used to evaluate patients' cardiac function and coronary heart disease symptoms, and Minnesota Heart Failure Quality of Life Questionnaire (MLHFQ) was used to evaluate the quality of life of patients with heart failure. The SF-36 health questionnaire was used to evaluate the overall health status and quality of life of patients.
angina pectoris readmission | From enrollment to the end of follow up at 5 years
heart failure | From enrollment to the end of follow up at 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No